CLINICAL TRIAL: NCT05196555
Title: Microscopic Surgical Repair of Cleft Palate With Inravelar Veloplasty
Brief Title: Cleft Palate With Intravelar Veloplasty Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Maxillo_2021
Record Dates: First submitted 2021-12-17; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- microscopic surgical repair of cleft palate with intravelar veloplasty (IVVP) (Experimental)
  Interventions: Procedure: Repair of cleft palate with intravelar veloplasty (IVVP)

INTERVENTIONS:
Procedure: Repair of cleft palate with intravelar veloplasty (IVVP) — A triangular flap is designed comprising new epithelial tissue which will be turned over to help close the nasal mucosa. Using a single hook, the oral mucosa and gland layer is separated from the muscle layer. Dissection of the greater palatine nerve-vessel bundle. The anterior palatal flap is raised by a curved elevator. The closure of the nasal mucosa and muscle is completed. Dissection of Velo Palatine Levator begins from the posterior rim of muscle and 5 mm from the midline.

SUMMARY:
Cleft palate repair is the most important component of cleft surgery, not only in that it determines the outcome as far as speech and communication are concerned, but also in that it potentially has the greatest impact on maxillary growth and the dental arch relationship. Sommerlad technique has been described as a more physiological approach, aiming to restore the anatomy of the velum. This technique, often described as radical intravelar veloplasty, has the following distinctive components: a radical retroposition of velar musculature (m. levator veli palatini, m. palatoglossus, and m. palatopharyngeus), combined with minimal dissection of the hard palate, a tensor tenotomy, and the repair of the m. levator sling

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated cleft palate age from 9 months to 18 years.
* Patients with submucous cleft.
* Velopharyngeal incompetence (VPI) for palatal re-repair.

Exclusion Criteria:

* Medically unfit patients.
* Syndromic patients with cleft lip and palate.
* Patients with cleft palate associated with multiple congenital anomalies.
* Patients with neurological disorders.

Ages: 9 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
change in soft palate elevation | Baseline, immediately after procedure
  Observing the range of motion of soft palate using videofluoroscopy
change in tongue motion assessment | Baseline, immediately after procedure
  Observing the range of tongue motion using videofluoroscopy
change in lips motion assessment | Baseline, immediately after procedure
  Observing the range of lips motion using videofluoroscopy
change in nasal airflow | Baseline, immediately after procedure
  Using Nasometer II model 6450 to assess the ratio of oral airflow to nasal airflow.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt